CLINICAL TRIAL: NCT01062711
Title: Responses of Muscle and Whole-body Protein Turnover to Ingestion of Differing Doses of Whey and Soy Protein With and Without Resistance Exercise in Elderly Men
Brief Title: Dose Response of Whey and Soy Protein Ingestion With and Without Resistance Exercise in Elderly Men
Acronym: NDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Stuart Phillips, Ph.D., Professor and Associate Chair, Graduate Studies, McMaster University, Department of Kinesiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DMI 1484
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Sarcopenia
Keywords: sarcopenia; muscle; protein; muscle protein synthesis; muscle protein breakdown; whey; soy; casein; dose response; resistance exercise; unilateral; knee extension; whole body protein
MeSH Terms: conditions — Sarcopenia | interventions — Whey; Soybean Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- Control group 0 g protein (Other): Control group in which a placebo drink containing no protein is given following unilateral knee extension exercise
  Interventions: Dietary Supplement: Whey or soy protein
- 10g whey (Experimental): 10g whey protein given following unilateral knee extension exercise
  Interventions: Dietary Supplement: Whey or soy protein
- 20g whey (Experimental): 20g whey protein given following unilateral knee extension exercise
  Interventions: Dietary Supplement: Whey or soy protein
- 30g whey (Experimental): 30g whey protein given following unilateral knee extension exercise
  Interventions: Dietary Supplement: Whey or soy protein
- 40g whey (Experimental): 40g whey protein given following unilateral knee extension exercise
  Interventions: Dietary Supplement: Whey or soy protein
- 20g soy (Experimental): 20g soy protein given following unilateral knee extension exercise
  Interventions: Dietary Supplement: Whey or soy protein
- 40g soy (Experimental): 40g soy protein given following unilateral knee extension exercise
  Interventions: Dietary Supplement: Whey or soy protein

INTERVENTIONS:
Dietary Supplement: Whey or soy protein — Whey and casein are isolated milk proteins

SUMMARY:
When we age, we lose muscle. It is not exactly clear why this happens, but we do know that this muscle loss can increase health risks and lead to health problems. Lifting weights (i.e. performing resistance exercise) and proper nutrition, in particular eating enough high quality protein, can help slow the loss of muscle mass or potentially even reverse it. Protein and resistance exercise are thought to do this by stimulating your muscle to make more proteins and/or potentially by slowing down the rate at which your body breaks proteins down. Whey protein is a high quality protein isolated from milk and is known to stimulate new protein synthesis for all proteins in your body. However, to date, the effect that whey protein has on muscle protein synthesis, particularly in the elderly has yet to be determined. Thus the purposes of this study are: 1) to determine if whey is an effective source of protein that will stimulate muscle protein synthesis in the elderly, similar to what we have previously seen in young persons; 2) to determine the smallest amount of whey protein to consume to maximally stimulate your muscle to make new proteins; 3) to see if performing resistance exercise will augment the increase in new muscle protein synthesis with whey consumption; and 4) to try and found out if whey is more effective than soy protein in stimulating new muscle protein synthesis and suppressing muscle protein breakdown in the elderly, similar to what we have previously seen in young persons

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 60 to 80 years old
* Non-smoker
* Generally healthy and can tolerate the resistance exercise and protein drink

Exclusion Criteria:

* Allergies to whey, casein or soy
* Health problems such as: heart disease, rheumatoid arthritis of the knee joint, diabetes, poor lung function, uncontrolled hypertension, or any health conditions that might put participants at risks for this study
* Failed clearance for exercise participation by their medical doctor
* Failed an exercise stress test
* Taking metformin and/or other medications for the control of blood glucose even though one might not be classified as diabetic
* Taking prescribed blood thinners such as warfarin and heparin but excluding aspirin
* Taking medications for lung and kidney conditions but excluding medication for asthma that is under control

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | Acute within the day
whole body amino acid oxidation | acute within the day

SECONDARY OUTCOMES:
muscle protein breakdown | Acute within the day
serum insulin | acute within the day
plasma amino acid concentrations | acute within the day

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Ph.D., Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada